CLINICAL TRIAL: NCT03125824
Title: Soliton Planar Acoustic Wave Device System for Dermal Tattoo Clearing Human Trial
Brief Title: Soliton Planar Acoustic Wave Device System for Dermal Tattoo Clearing Human Trial Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soliton (Industry)
Collaborators: MedSource LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soliton 2017-001
Record Dates: First submitted 2017-04-06; First posted 2017-04-24 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Tattooing

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Tattoos previously treated in Soliton 2016-001 trial (Other): Identical tattoos treated by Laser + AWD in Soliton's previous trial
  Interventions: Device: Soliton Acoustic Wave Device

INTERVENTIONS:
Device: Soliton Acoustic Wave Device — Treatment of tattoos with Soliton Acoustic Wave Device as an accessory to laser
  Other Names: AWD

SUMMARY:
To further evaluate accelerated fading resulting from additional treatment sessions of Soliton AWD as accessory to laser in tattoo reduction treatment.

DETAILED DESCRIPTION:
To further evaluate accelerated fading resulting from additional treatment sessions of multi-pass Q-Switched laser with the Soliton Planar Acoustic Wave Device System (AWD) as an accessory to Q-Switched laser in tattoo reduction treatment.

ELIGIBILITY:
Inclusion Criteria:

* Range of Fitzpatrick skin color scores I to III
* The identical tattoo located on the arms, legs, and torso treated by Q-Switched laser and Laser + AWD during Soliton's previous 2016-001 clinical trial
* Black ink only. Other ink colors may be present, but areas of black only tattoo should meet inclusion criteria
* Approximately 1" x 3" tattoo with at least 30-50% of the treatment area containing black tattoo ink

Exclusion Criteria:

* Subject is pregnant or planning to become pregnant during the duration of the study
* Medical disorder that would hinder the wound healing or immune response (no blood disorder, diabetes, inflammatory disease, etc.)
* Skin disorders (skin infections or rashes, scarring, moles,birthmarks, psoriasis, etc.)
* Any surgical procedure in the prior 3 months, or planned during the duration of the study
* Active electronic implants such as pacemakers, defibrillators, cochlear implants, nerve/brain stimulators, etc.
* Moderate to heavy tanning on and around the tattoo to be treated as determined by the Principle Investigator.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Tattoo clearance | 12 weeks
  To evaluate changes in accelerated fading of previously treated tattoos from original treatment with additional treatment sessions of Soliton Acoustic Wave Device as an accessory to laser treatment through comparison of photographic evidence. Changes are measured by comparing photos of the tattoos after the original treatment to photos of the tattoos after additional treatment.

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events for Safety Reporting | 12 weeks
  Adverse Events and complications evaluated for severity and device relationship

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cappelli, MD, Study Director — Soliton
Locations (1):
- SkinCare Physicians, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No